CLINICAL TRIAL: NCT04608032
Title: Neuropsychological Assessment of Remediation for Cognitive Impairments in Schizophrenia
Acronym: NARCIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Clémence ISAAC, Principal Investigator, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10477M-NARCIS
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenia; Neurocognition; Social cognition; Metacognition; Cognitive remediation
MeSH Terms: conditions — Schizophrenia | interventions — Thor protein, Drosophila

STUDY DESIGN:
Intervention Model Description: The first group is about cognitive remediation therapy (ECo-Sz). The second group is about recovery oriented therapy (ThOR).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ecological Cognitive training program for schizophrenia spectrum disorder [ECo-Sz] (Experimental): To inform the patient about cognitive impairments and their repercussions ; to train the patient in problem-solving skills through exercices ; to implement strategies in daily life. Duration : two month. Frequency : Two one hour individual sessions and one hour of at-home training per week. Modalities : pen and papers exercices (tools, token, cards, maps and chessboard). Modules : Psychoeducation, Attention, Memory, Executive functions, Social cognition and metacognition, Functional impairments
  Interventions: Other: [Eco-Sz] Ecological Cognitive training program for schizophrenia spectrum disorder
- [THoR] Recovery-Oriented Therapy (Active Comparator): Individual psychotherapy sessions focussing on autonomy in daily life, management of mood disorders' and functional impact, social skills, motivation and the regulation of sleep and daily activities
  Interventions: Other: Recovery-Oriented Therapy

INTERVENTIONS:
Other: [Eco-Sz] Ecological Cognitive training program for schizophrenia spectrum disorder — The first group will have [Eco-Sz] Ecological Cognitive training program for schizophrenia spectrum disorder
  Other Names: [Eco-Sz]
  Arms: Ecological Cognitive training program for schizophrenia spectrum disorder [ECo-Sz]
Other: Recovery-Oriented Therapy — The second group will have [THoR] Recovery-Oriented Therapy
  Other Names: [THoR]
  Arms: [THoR] Recovery-Oriented Therapy

SUMMARY:
This study evaluates the effect of a cognitive remediation program on neurocognitive, social cognitive and metacognitive functions designed for patients living with a schizophrenia spectrum disorder.

DETAILED DESCRIPTION:
Evaluation of the specific therapeutic efficacy of the ecological cognitive remediation program for schizophrenia spectrum disorder [ECo-Sz] on neurocognitive deficits, social cognition deficits and metacognition deficits of patients with a schizophrenia spectrum disorder.

In this double-blind (patients, outcomes assessors) controlled randomized trial the investigators compare patients receiving Ecological Cognitive training program for schizophrenia spectrum disorder [ECo-Sz] to patients benefiting from recovery-oriented therapy [ThOR]. Patients are treated for two months and monitored for four months.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia Disorder diagnosis, according to Diagnostic and Statistical Manual of mental disorders - Fifth edition (DSM-V) - Patient stabilized in terms of positive and negative symptomatology (absence or presence of weak positive and negative symptoms)
* Positive and Negative stable symptoms (no or few positive and negative symptoms)
* Stable and effective minimum dose of medication (antipsychotic) for the last three months
* Cognitive complaint expressed by the patient
* Informed consent form read, initialed and signed
* Understanding of spoken and read French
* Patient registered on the social welfare system

Exclusion Criteria:

* Other diagnosis at the forefront than Schizophrenia of the DSM-V
* Medical history neurological disorder resulting in hospitalization
* Acute episode in the last three month
* Somatic disorders resulting in cognitive impairment
* Engagement in a research protocol either currently or over the last month
* Neuropsychological assessment evaluation during the last six month
* Patients under the protection of a conservator (simple or reinforced)
* Individuals in vulnerable circumstances

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
STROOP | pre-inclusion
  Interference score
TMTB | pre-inclusion
  Trail Making Test
Litteral score of Verbal fluences | pre-inclusion
  Litteral score of Verbal fluences
GO/NOGO | pre-inclusion
  cognitive control score
tower of Hanoi | pre-inclusion
  Tower planning total score from tower of Hanoi
Matrix test (WAIS-IV) | pre-inclusion
  The perceptual reasoning score of the Matrix test.

SECONDARY OUTCOMES:
Mini-500 | pre-inclusion
  (Entretien structuré Neuropsychiatrique International
CTQ | pre-inclusion
  Childhood Trauma Questionnaire - minimum value = 28 - maximum value = 112
PANSS | pre-inclusion
  Positive and Negative Syndrome Scale - minimum value = 30 - maximum value = 210
EESEP | Eighteen week
  Self-Efficacity Rating Scale - minimum value = 21 - maximum value = 105
EESEP | Twenty six week
  Self-Efficacity Rating Scale - minimum value = 21 - maximum value = 105
ERF | First week
  Functional Impact Scale - minimum value = 5 - maximum value = 35
ERF | Ten week
  Functional Impact Scale - minimum value = 5 - maximum value = 35
ERF | Eighteen week
  Functional Impact Scale - minimum value = 5 - maximum value = 35
ERF | Twenty six week
  Functional Impact Scale - minimum value = 5 - maximum value = 35
ERF-CS | First week
  Functional Impact Scale for Social Cognition disorders- minimum value = 4 - maximum value = 20
ERF-CS | Ten week
  Functional Impact Scale for Social Cognition disorders- minimum value = 4 - maximum value = 20
ERF-CS | Eighteen week
  Functional Impact Scale for Social Cognition disorders- minimum value = 4 - maximum value = 20
ERF-CS | Twenty six week
  Functional Impact Scale for Social Cognition disorders- minimum value = 4 - maximum value = 20
MCQ-30 | First week
  Short French Meta-Cognitions Questionnaire - minimum value = 30 - maximum value = 120
MCQ-30 | Ten week
  Short French Meta-Cognitions Questionnaire - minimum value = 30 - maximum value = 120
MCQ-30 | Eighteen week
  Short French Meta-Cognitions Questionnaire - minimum value = 30 - maximum value = 120
MCQ-30 | Twenty six week
  Short French Meta-Cognitions Questionnaire - minimum value = 30 - maximum value = 120
QFS | First week
  Social Functioning Questionnaire - no minimum or maximum value
QFS | Ten week
  Social Functioning Questionnaire - no minimum or maximum value
QFS | Eighteen week
  Social Functioning Questionnaire - no minimum or maximum value
QFS | Twenty six week
  Social Functioning Questionnaire - no minimum or maximum value
SAIQ | First week
  Self-Appraisal of Illness Questionnaire - minimum value = 17- maximum value = 68
SAIQ | Ten week
  Self-Appraisal of Illness Questionnaire - minimum value = 17- maximum value = 68
SAIQ | Eighteen week
  Self-Appraisal of Illness Questionnaire - minimum value = 17- maximum value = 68
SAIQ | Twenty six week
  Self-Appraisal of Illness Questionnaire - minimum value = 17- maximum value = 68
SCS | First week
  Revised Self-Consciousness Scale - minimum value = 0 - maximum value = 66
SCS | Ten week
  Revised Self-Consciousness Scale- minimum value = 0 - maximum value = 66
SCS | Eighteen week
  Revised Self-Consciousness Scale - minimum value = 0 - maximum value = 66
SCS | Twenty six week
  Revised Self-Consciousness Scale - minimum value = 0 - maximum value = 66
SDS | First week
  Social Desirability Scale - minimum value = 0 - maximum value = 33
SDS | Ten week
  Social Desirability Scale - minimum value = 0 - maximum value = 33
SDS | Eighteen week
  Social Desirability Scale - minimum value = 0 - maximum value = 33
SDS | Twenty six week
  Social Desirability Scale - minimum value = 0 - maximum value = 33
STORI | First week
  Stage of Recovery Instrument - minimum value = 0 - maximum value = 50
STORI | Ten week
  Stage of Recovery Instrument - minimum value = 0 - maximum value = 50
STORI | Eighteen week
  Stage of Recovery Instrument - minimum value = 0 - maximum value = 50
STORI | Twenty six week
  Stage of Recovery Instrument - minimum value = 0 - maximum value = 50

OTHER OUTCOMES:
FAUX-PAS Test | First week
  A test assessing first and second degree theory of mind through short stories and pictures involved two or three characters - minimum value = 0 - maximum value = 60
FAUX-PAS Test | Ten week week
  A test assessing first and second degree theory of mind through short stories and pictures involved two or three characters - minimum value = 0 - maximum value = 60
FAUX-PAS Test | Eighteen week week
  A test assessing first and second degree theory of mind through short stories and pictures involved two or three characters - minimum value = 0 - maximum value = 60
FAUX-PAS Test | Twenty six week
  A test assessing first and second degree theory of mind through short stories and pictures involved two or three characters - minimum value = 0 - maximum value = 60
The Rey/Taylor complex figure test | First week
  The test is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by ping it freehand and then drawing from memory. This test permits the evaluation of visuospatial abilities, memory, attention, planning and working memory - minimum value = 0 - maximum value = 36
The Rey/Taylor complex figure test | Ten week
  The test is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by ping it freehand and then drawing from memory. This test permits the evaluation of visuospatial abilities, memory, attention, planning and working memory - minimum value = 0 - maximum value = 36
The Rey/Taylor complex figure test | Eighteen week
  The test is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by ping it freehand and then drawing from memory. This test permits the evaluation of visuospatial abilities, memory, attention, planning and working memory - minimum value = 0 - maximum value = 36
The Rey/Taylor complex figure test | Twenty six week
  The test is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing, first by ping it freehand and then drawing from memory. This test permits the evaluation of visuospatial abilities, memory, attention, planning and working memory - minimum value = 0 - maximum value = 36
MEM IV Logical Memory | First week
  Composite score of the Weschler Memory Scale - fourth edition
MEM IV Logical Memory | Ten week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Logical Memory | Eighteen week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Logical Memory | Twenty six week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Symbol Memory | First week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Symbol Memory | Ten week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Symbol Memory | Eighteen week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
MEM IV Symbol Memory | Twenty six week
  Composite score of the Weschler Memory Scale - fourth edition - minimum value = 0 - maximum value = 20
The Balloon Analogue Risk Task | First week
  The Balloon Analogue Risk Task is a computerized measure of risk taking behavior - no minimum or maximum value
The Balloon Analogue Risk Task | Ten week
  The Balloon Analogue Risk Task is a computerized measure of risk taking behavior - no minimum or maximum value
The Balloon Analogue Risk Task | Eighteen week
  The Balloon Analogue Risk Task is a computerized measure of risk taking behavior - no minimum or maximum value
The Balloon Analogue Risk Task | Twenty six week
  The Balloon Analogue Risk Task is a computerized measure of risk taking behavior - no minimum or maximum value
D2 Test | First week
  The test is neuropsychological measure of selective and sustained attention and visual scanning speed - no minimum or maximum value
D2 Test | Ten week
  The test is neuropsychological measure of selective and sustained attention and visual scanning speed - no minimum or maximum value
D2 Test | Eighteen week
  The test is neuropsychological measure of selective and sustained attention and visual scanning speed - no minimum or maximum value
D2 Test | Twenty six week
  The test is neuropsychological measure of selective and sustained attention and visual scanning speed - no minimum or maximum value
ToM-15 | First week
  The test is a task assessing theory of mind abilities you cannot move more than one disk at a time; a disk can only be placed on another disk larger than it or on an empty location - no minimum or maximum value
ToM-15 | Ten week
  The test is a task assessing theory of mind abilities you cannot move more than one disk at a time; a disk can only be placed on another disk larger than it or on an empty location - no minimum or maximum value
ToM-15 | Eighteen week
  The test is a task assessing theory of mind abilities you cannot move more than one disk at a time; a disk can only be placed on another disk larger than it or on an empty location - no minimum or maximum value
ToM-15 | Twenty six week
  The test is a task assessing theory of mind abilities you cannot move more than one disk at a time; a disk can only be placed on another disk larger than it or on an empty location - no minimum or maximum value
Cubes Subtest | First week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Cubes Subtest | Ten week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Cubes Subtest | Eighteen week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Cubes Subtest | Twenty six week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Visual Puzzle Subtest | First week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Visual Puzzle Subtest | Ten week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Visual Puzzle Subtest | Eighteen week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Visual Puzzle Subtest | Twenty six week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Similiraties Subtest | First week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Similiraties Subtest | Ten week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Similiraties Subtest | Eighteen week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Similiraties Subtest | Twenty six week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Working Memory Subtest | First week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Working Memory Subtest | Ten week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Working Memory Subtest | Eighteen week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20
Working Memory Subtest | Twenty six week
  Composite score of Weschler Adult Intelligence Scale - fourth edition - minimum value = 0 - maximum value = 20

CONTACTS AND LOCATIONS:
Overall Officials: Clémence ISAAC, PHD, Principal Investigator — URC EPS Ville Evrard
Locations (2):
- France (2):
  - Ch Ville Evrard, Neuilly-sur-Marne
  - URC Ville Evrard, Neuilly-sur-Marne

IPD SHARING:
Plan to Share IPD: No